CLINICAL TRIAL: NCT02108561
Title: Does Breast Tumor Heterogeneity Necessitate Additional HER2 Testing on the Surgical Specimens?
Brief Title: Breast Cancer Tumor Heterogeneity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Anne Arundel Health System Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 505185
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Heterogeneity Her2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer: Post Surgical Her2 testing
  Interventions: Other: Post Surgical Her2 testing

INTERVENTIONS:
Other: Post Surgical Her2 testing — Eligible patients will have post surgical Her2 testing on the primary tumor, a satellite lesion and a tumor positive node. The results will be provided to medical oncologist, who will comment as to whether the additional testing will prompt treatment recommendation changes

SUMMARY:
Breast cancer biomarkers are usually performed on core needle biopsy (CNB) specimens and are not routinely repeated on surgical specimens (SS). However, preliminary data suggests that testing these biomarkers, on SS when compared to CNB samples can lead to different results. Our hypothesis is that The aim of this study is to identify a group of women with invasive breast cancer who may benefit from additional HER2 testing on their SS to ensure that areas of HER2 amplification are not missed. Another aim is to determine whether further HER2 testing on the SS in select patients would lead to changes in breast cancer treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Women > age 18 with capacity to consent
2. Invasive breast cancer identified on CNB at AAMC within 45 days of study consent
3. IHC biomarkers performed on original CNB (including HER2)
4. Tumors with greater than 2cm of invasive disease (measured radiographically prior to resection or microscopically after resection), or
5. Multifocal or multicentric tumors

Exclusion Criteria:

1. Men
2. Women with HER2 positive tumors detected on CNB specimens
3. Women receiving neoadjuvant chemotherapy
4. Women whose CNB or surgical resection was performed at a hospital other than AAMC. If the CNB prior to resection was repeated at AAMC and new tumor biomarkers were performed, then the patient is eligible for enrollment
5. Women whose IHC marker results were inconclusive on CNB or not performed -

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer pre-surgical patients
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12-22 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Benefit of additional Her2 testing | 2 years
  To identify a subset of women with invasive breast cancer who may benefit from additional Her2 testing (by immunochemistry and FISH) on their surgical specimen to ensure that areas of Her2 amplification are not missed due to sampling error of the core needle biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States